CLINICAL TRIAL: NCT05429554
Title: The Impact of Metformin and Dipeptidyl Peptidase- 4 Inhibitors on Cognitive Function and Cardiovascular Protection in Type 2 Diabetic Patients
Brief Title: The Effect of Metformin and DPP4 Inhibitors on Cognition and Cardiovascular Protection in Type 2 Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MTI University (Other)
Collaborators: National Institute of Diabetes and Endocrinology, Egypt (Unknown)
Responsible Party: Principal Investigator, Toka Hesham, Teaching assistant of Clinical Pharmacy, MTI University
Other Study IDs: IDEoo281
Record Dates: First submitted 2022-06-19; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group 1: patients will be treated with DPP4 inhibitor + metformin
  Interventions: Drug: Vildagliptin
- control: patients will be treated with metformin without DPP4 inhibitor.

INTERVENTIONS:
Drug: Vildagliptin — observe the effect of vildagliptin on cognitive function and cardiovascular in diabetic patients
  Groups: group 1

SUMMARY:
The Impact of Metformin and Dipeptidyl Peptidase- 4 Inhibitors on Cognitive Function and cardiovascular protection in Type 2 Diabetic Patients

DETAILED DESCRIPTION:
This study aims to investigate the effect of daily oral DPP4 inhibitors and oral metformin on neurodegeneration in type 2 diabetic patients.

This study aims to compare between the cardiovascular protective properties of DPP-4 inhibitors and Metformin in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient should be diagnosed with Type 2 diabetes mellitus (T2DM) and guided with HA1c ≥7, age ≥40 years.
* moderate hypertension.

Exclusion Criteria:

* • Diabetic patients who have been currently receiving anti-diabetic agents other than metformin and/or insulin

  * Patients with type 1 DM, active liver disease, recent history of cardiovascular disease (acute coronary syndrome, coronary artery intervention, New York Heart Association Class III/IV heart failure, stroke, transient ischemic neurologic event, or new/worsening symptoms of coronary heart disease or cerebrovascular disease), severe peripheral vascular disease, triglyceride levels ≥ 600 mg/dL, history of HIV infection, pancreatitis, malignancy or clinically important hematologic disorder, and an estimated glomerular filtration rate (eGFR; calculated using the Modification of Diet in Renal Disease formula) less than 30 mL/min/1.73 m2.
  * Moreover, patients with dementia, AD, those were in delirium status during evaluation period, patients with psychotic disease (schizoaffective disorder, etc.)
  * Alcohol and substance addiction were not enrolled in the study.
  * Also, patients who have any hypersensitivity to metformin or to DPP4 inhibitors were also excluded.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study contains 2 groups each group consists of 30 patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
improve the neurodegeneration and cardiovascular effect in diabetic patients | September 2022
  improve the cognition and cardiovascular effect in type 2 diabetic patients

CONTACTS AND LOCATIONS:
Overall Officials: Toka Hesham, Principal Investigator — Bachelor of Pharmacy and Pharmaceutical sciences (Clinical Pharmacy)
Locations (1):
- National Institute of diabetes and endocrinology, Cairo, Al Kasr Al Aini, Egypt